CLINICAL TRIAL: NCT06866769
Title: Comparación De La Eficacia Entre Biomarcadores Y Ecografía Con Contraste Frente a Angio-TC En El Seguimiento De Aneurismas De Aorta Abdominal (AAA) Tras Reparación Endovascular (EVAR)
Brief Title: Efficacy of Biomarkers and CEUS Versus CTA in AAA Follow-up Post-EVAR
Acronym: EVAR-markers
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: EVAR
Record Dates: First submitted 2025-01-24; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture
Keywords: Abdominal Aortic Aneurysm (AAA); Endovascular Aneurysm Repair (EVAR); Contrast-enhanced ultrasound (CEUS); Computed tomography angiography (CTA); Biomarkers.
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study cohort: Inclusion Criteria:
  * patients with AAA under follow-up who are going to be treated with EVAR.
  * signed informed consent to perform CTA, CEUS and for the determination of biomarkers.
  Exclusion Criteria:
  * patients with inflammatory abdominal aortic aneurysms or ruptured aneurysm.
  Interventions: Diagnostic Test: CTA

INTERVENTIONS:
Diagnostic Test: CTA — The levels of biomarkers are determined before (within 30 days prior to the procedure) and after the implantation of the stent (24-48 hours, 1 month, 3 months, 6 months, and at 1 year), along with the performance of a contrast-enhanced ultrasound. Additionally, a follow-up CT angiography is performed to validate the concordance, that is, to assess if there are changes in the biomarker values determined one month after the implantation of the stent compared to the baseline values that may suggest the presence of complications (endoleaks, infection, thrombosis, etc.).
  Other Names: Ultrasound image enhancement

SUMMARY:
This prospective observational study evaluates the efficacy of contrast-enhanced ultrasound and biomarker determination in the follow-up of patients with abdominal aortic aneurysm (AAA) treated with Endovascular Aneurysm Repair (EVAR). Currently, computed tomography angiography (CTA) is the standard for follow-up, although it has disadvantages such as radiation exposure and the use of iodinated contrasts. Contrast-enhanced ultrasound (CEUS), free of radiation and nephrotoxicity, and biomarkers could reduce the need for CTA minimizing the associated risks. Biomarkers will be measured before and after EVAR and CEUS will be performed at various time points and compared with CTA results to validate concordance and effectiveness in detecting endoleaks and aneurysm remodeling. The objectives include determining the efficacy of these combined methods and establishing a follow-up protocol that reduces exposure to radiation and iodinated contrast agents.

DETAILED DESCRIPTION:
Background/Rationale:

Patients with AAA who have undergone EVAR of the abdominal aortic aneurysm require indefinite follow-up since a 4-year complication rate after EVAR of up to 40% has been described in some series.

In some patients a decrease in the diameters of the residual aneurysm sac after EVAR has been described, which is known as remodeling.

CTA is the gold standard imaging technique for the follow-up of these patients, although it has the disadvantage of using ionizing radiation and iodinated contrasts that are nephrotoxic and can produce hypersensitivity reactions. Furthermore, there is no consensus on which protocol is the most suitable (one phase, two phases or three phases). Currently, in our hospital, three-phase CTA is being performed, as well as CTA with the Split Bolus technique, which allows the acquisition of images in arterial and venous phases in a single acquisition, thus reducing radiation doses; a correlation between both techniques of 85.7-100% and a decrease in radiation doses of between 30-78% has been described.

An alternative to CTA is CEUS that presents a sensitivity of 90.5% (22-100%) and a specificity of 90.65% (71-100%) for the detection of endoleaks. It is a technique that does not use ionizing radiation; furthermore, ultrasound contrasts are not nephrotoxic and hypersensitivity reactions to them are exceptional. In addition, there are publications concerning the determination of biomarkers in the follow-up of patients with AAA both before and after treatment with EVAR.

Hypothesis:

Performing CEUS together with biomarker determination in patients with AAA treated by EVAR would allow reducing the number of CTA to these patients; and, therefore, radiation doses and the use of iodinated contrasts that may cause nephrotoxicity, as well as hypersensitivity reactions.

Primary objectives:

1. - To determine whether the combination of biomarker levels together with CEUS in the follow-up of treated AAA patients is as effective as performing CTA to detect endoleaks.
2. - To validate the usefulness of CEUS together with biomarker determination in the follow-up of these patients.

Secondary Objectives:

1.- To determine the cost-effectiveness of biomarkers in the follow-up of these patients.

To establish a protocol for the follow-up of patients with AAA treated with EVAR, including biomarkers and CEUS.

3.-To reduce radiation doses in the follow-up of patients with AAA treated with EVAR.

Methodology:

Prospective observational study. Biomarker levels will be determined before (within 30 days prior to the procedure) and after stent implantation (24-48 h, 1 month, 3 months, 6 months and 1 year) together with contrast echography. In addition, a control CTA will be performed to validate concordance. These biomarkers will be analyzed comparing the values obtained in patients with endoleaks versus patients without endoleaks, as well as in those with aneurysm remodeling.

ELIGIBILITY:
Inclusion Criteria:

* patients with AAA under follow-up who are going to be treated with EVAR.
* signed informed consent to perform CTA, CEUS and for the determination of biomarkers.

Exclusion Criteria:

* patients with inflammatory abdominal aortic aneurysms or ruptured aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AAA treated with EVAR will undergo a clinical evaluation prior to the procedure, assessing inclusion and exclusion criteria. A determination of biomarkers will be carried out to determine their values before the procedure, which will be carried out within 30 days of said assessment. Patients who meet the inclusion criteria will be studied prospectively to assess the effectiveness of biomarker levels along with CEUS to detect endoleaks.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Biomarkers Levels for Endoleak Detection Post-EVAR Treatment | Biomarkers will be evaluated before (within 30 days prior to the procedure) and after implantation of the endoprosthesis (24-48 hours, 1 month, 3 months, 6 months, and 1 year).
  To determine if biomarker levels can detect endoleaks as a complication in patients treated for AAA, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Endoleak Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Extracellular Matrix Remodeling Markers: Matrix Metalloproteinase-9 (MMP-9) (ng/mL)
  * Renal Function Markers: Cystatin C (mg/L)
  * Coagulation Markers: von Willebrand Factor (%), Factor VIII (IU/dL)
  Analysis: Each biomarker will be grouped into clinically relevant categories and analyzed as an independent measure within its respective category to assess its correlation with endoleak occurrence.
Biomarkers Levels for Thrombosis Detection Post-EVAR Treatment | Biomarkers will be evaluated before (within 30 days prior to the procedure) and after implantation of the endoprosthesis (24-48 hours, 1 month, 3 months, 6 months, and 1 year).
  To determine if biomarker levels detect thrombosis in AAA patients, changes will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Thrombosis Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Coagulation Markers: Prothrombin Time (PT) (seconds), Activated Partial Thromboplastin Time (aPTT) (seconds), Derived Fibrinogen (mg/dL), Factor XIII (%)
  * Platelet Function Markers: PFA-100 COL/ADP (seconds), PFA-100 COL/EPI (seconds)
  * Anticoagulation Markers: Protein C (%), Protein S (%), Antithrombin (%)
  * Thrombophilia Markers: Lupus Anticoagulant (Presence/Absence), Activated Protein C Resistance ((+/-)), Prothrombin G20210A Mutation ((+/-)), Factor V Leiden Mutation (G1691A) ((+/-))
  Analysis: Each biomarker will be grouped into clinically relevant categories and analyzed as an independent measure within its respective category to track changes and assess their correlation with thrombosis.
Biomarkers Levels for Infection Detection Post-EVAR Treatment | Biomarkers will be evaluated before (within 30 days prior to the procedure) and after implantation of the endoprosthesis (24-48 hours, 1 month, 3 months, 6 months, and 1 year).
  To determine if biomarker levels can detect infection as a complication in patients treated for AAA, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Infection Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  - Inflammatory Markers: C-Reactive Protein (CRP) (mg/L); Procalcitonin (ng/mL); IL-6 (pg/mL); IL-8 (pg/mL); TNF-α (pg/mL); Serum Calprotectin (µg/mL)
  Analysis: Each biomarker will be grouped as an inflammatory marker and analyzed as an independent measure to track changes and assess its correlation with infection.
Biomarker Levels for Prosthesis-Related Complication Detection Post-EVAR Treatment | Biomarkers will be evaluated before (within 30 days prior to the procedure) and after implantation of the endoprosthesis (24-48 hours, 1 month, 3 months, 6 months, and 1 year).
  To determine whether biomarker levels can detect complications such as displacement, dislocation, and plication of the prosthesis in patients treated for AAA, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Biomarkers Related to Prosthesis Issues from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Lipid Metabolism Markers: Apolipoprotein A1 (ApoA1) (mg/dL), Apolipoprotein B (ApoB) (mg/dL)
  * Hematological Markers: Reticulocytes (10³/mL)
  * Coagulation Markers: Quick Index (%)
  * Autoimmune Markers: Anticardiolipin Antibodies (IgG/IgM) (GPL/MPL units)
  Analysis: Each biomarker will be grouped into clinically relevant categories and treated as an independent measure within its respective category.
CEUS (Contrast-Enhanced Ultrasound) for Endoleak Detection Post-EVAR treatment | CEUS will be performed at baseline (within 30 days before the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  Objective: To determine if CEUS can detect endoleaks, thrombosis, infection, and complications related to protesis placement (displacement/dislocation of the prosthesis, plication of the prosthesis) in patients treated for AAA.
  • Units of Measure: Presence/absence of endoleaks, thrombosis, infection, displacement/dislocation of the prosthesis, plication of the prosthesis
  Comments: The presence or absence of endoleaks and other complications will be assessed, along with severity when applicable
Validation of CEUS for Endoleak and Complication Detection Post-EVAR treatment | CEUS will be performed at baseline (within 30 days before the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  Objective: To validate the use of Contrast-Enhanced Ultrasound (CEUS) for detecting endoleaks, thrombosis, infection, and complications related to protesis placement (displacement/dislocation of the prosthesis, plication of the prosthesis) in patients treated for AAA, compared to angio-CT (gold standard).
  * Units of Measure: Presence/absence of endoleaks, thrombosis, infection, displacement/dislocation of the prosthesis, plication of the prosthesis
  * Comparison Standard: Angio-CT (gold standard)
  Comments: The presence or absence of endoleaks and other complications will be assessed, along with severity when applicable. CEUS results will be compared to the angio-CT results for validation.
Validation of Biomarkers for Endoleaks Detection Post EVAR | Biomarkers will be assessed at baseline (within 30 days prior to the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  To validate biomarkers for detecting endoleaks as a post-EVAR complication, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Endoleak Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Extracellular Matrix Remodeling Markers: Matrix Metalloproteinase-9 (MMP-9) (ng/mL)
  * Renal Function Markers: Cystatin C (mg/L)
  * Coagulation Markers: von Willebrand Factor (%), Factor VIII (IU/dL)
  Analysis: Each biomarker will be grouped into clinically relevant categories and analyzed as an independent measure within its respective category to assess its correlation with endoleak occurrence
Validation of Biomarkers for Thrombosis Detection Post-EVAR treatment | Biomarkers will be assessed at baseline (within 30 days prior to the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  To validate biomarkers for detecting thrombosis as a post-EVAR complication, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Thrombosis Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Coagulation Markers: Prothrombin Time (PT) (seconds), Activated Partial Thromboplastin Time (aPTT) (seconds), Derived Fibrinogen (mg/dL), Factor XIII (%)
  * Platelet Function Markers: PFA-100 COL/ADP (seconds), PFA-100 COL/EPI (seconds)
  * Anticoagulation Markers: Protein C (%), Protein S (%), Antithrombin (%)
  * Thrombophilia Markers: Lupus Anticoagulant (Presence/Absence), Activated Protein C Resistance ((+/-)), Prothrombin G20210A Mutation ((+/-)), Factor V Leiden Mutation (G1691A) ((+/-))
  Analysis: Each biomarker will be grouped into clinically relevant categories and analyzed as an independent measure within its respective category to track changes and assess their correlation with thrombosis.
Validation of Biomarkers for Infection Detection Post-EVAR treatment | Biomarkers will be assessed at baseline (within 30 days prior to the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  To validate biomarkers for detecting infection as a post-EVAR complication, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Infection Biomarkers from baseline to 1 year.
  Biomarkers and Units of Measure:
  - Inflammatory Markers: C-Reactive Protein (CRP) (mg/L); Procalcitonin (ng/mL); IL-6 (pg/mL); IL-8 (pg/mL); TNF-α (pg/mL); Serum Calprotectin (µg/mL)
  Analysis: Each biomarker will be grouped as an inflammatory marker and analyzed as an independent measure to track changes and assess its correlation with infection.
Validation of Biomarkers for Prosthesis-Related Complication Detection Post-EVAR Treatment | Biomarkers will be assessed at baseline (within 30 days prior to the procedure) and after implantation of the endoprosthesis: 24-48 hours, 1 month, 3 months, 6 months, and 1 year.
  To validate biomarkers for detecting complications such as displacement, dislocation, and plication of the prosthesis, changes in biomarker levels will be compared to baseline values and subsequent assessments.
  Outcome Measure: Change in Biomarkers Related to Prosthesis Issues from baseline to 1 year.
  Biomarkers and Units of Measure:
  * Lipid Metabolism Markers: Apolipoprotein A1 (ApoA1) (mg/dL), Apolipoprotein B (ApoB) (mg/dL)
  * Hematological Markers: Reticulocytes (10³/mL)
  * Coagulation Markers: Quick Index (%)
  * Autoimmune Markers: Anticardiolipin Antibodies (IgG/IgM) (GPL/MPL units)
  Analysis: Each biomarker will be grouped into clinically relevant categories and analyzed as an independent measure within its respective category.

SECONDARY OUTCOMES:
Cost-Effectiveness of Biomarker Measurements in AAA Follow-Up Post-EVAR treatment | Biomarkers will be evaluated before (within 30 days prior to the procedure) and after implantation of the endoprosthesis (24-48 hours, 1 month, 3 months, 6 months, and 1 year).
  Objective: To evaluate the cost-effectiveness of biomarker determination in the follow-up of AAA patients treated with EVAR, using a Health Economic Evaluation framework.
  * Units of Measure: Cost of biomarker tests (in euros).
  * Analysis Method: Cost-Effectiveness Analysis (CEA) and Cost-Minimization Analysis (CMA).
  Comments: The cost-effectiveness analysis will compare the costs of biomarker measurements to clinical outcomes such as detection and management of complications.
Cost-Effectiveness of Imaging (CEUS and CTA) in AAA Follow-Up Post-EVAR treatment | Imaging techniques (CEUS and CTA) will be performed at the same time points as biomarker assessments (within 30 days before the procedure, and after implantation: 24-48 hours, 1 month, 3 months, 6 months, and 1 year)
  Objective: To evaluate the cost-effectiveness of imaging techniques (CEUS and CTA) for follow-up of AAA patients treated with EVAR.
  * Units of Measure: Cost per imaging session (in euros).
  * Analysis Method: Cost-Effectiveness Analysis (CEA) and Cost-Minimization Analysis (CMA).
  Comments: The cost-effectiveness of CEUS and CTA will be assessed in relation to clinical outcomes, like the detection and management of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Sanchís García, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No